CLINICAL TRIAL: NCT05789134
Title: Mycoplasma Genitalium Infection and Associated Antimicrobial Resistance Among HIV-infected Male in Hong Kong
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Ngai Sze WONG, Assistant Professor, Chinese University of Hong Kong
Other Study IDs: 22210282
Record Dates: First submitted 2023-03-16; First posted 2023-03-29 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: STI; Mycoplasma Genitalium Infection
Keywords: chlamydia trachomatis; Mycoplasma Genitalium Infection; Neisseria gonorrhoeae; men who have sex with men; heterosexual men; people living with HIV
MeSH Terms: conditions — Sexually Transmitted Diseases; Homosexuality

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — urine specimen, rectal swab, pharyngeal swab
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: self-sampling kits for STI testing in the laboratory — Participants will receive the self-sampling kits and their submitted samples would be sent to laboratory for testing

SUMMARY:
Worldwide, Mycoplasma genitalium (MG) is increasingly reported as an emerging cause of sexually transmitted infections. Internationally, the prevalence of MG is higher in male with urethritis and community groups especially among people living with HIV (PLHIV). While MG is treatable, antimicrobial resistance is a rising concern. This cross-sectional study aims to determine the prevalence of MG infection and the antimicrobial resistance pattern in HIV-infected male in Hong Kong.

A total of 750 HIV-infected male attending HIV specialist clinic in Hong Kong would be recruited. The main outcome measures include prevalence of MG and resistance mutations to macrolide/fluoroquinolone in HIV-infected male; prevalence of MG/STI co-infections, as defined by concurrent detection of MG and one or more other bacterial STI.

DETAILED DESCRIPTION:
A total of 750 HIV-infected male attending HIV specialist clinic in Hong Kong would be recruited. An online questionnaire would be self-administered. The participants would self-collect urine sample, rectal and pharyngeal swabs for MG, Chlamydia trachomatis (CT) and Neisseria Gonorrhoeae (NG) screening by nucleic acid amplification tests, and MG genotypic resistance mutations detection. Clinical data would be transcribed from medical records of recruited subjects.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 or older, male, HIV-infected, and are attendees of the HIV specialist clinic, and can communicate in written and spoken English or Chinese

Exclusion Criteria:

* not able to provide consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: HIV-infected male who are attending the HIV specialist clinic in Hong Kong
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2023-07-24 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
prevalence of MG infection | 1 year
  detection of MG infections in self-collected samples divided by the total number of samples collected
prevalence of MG resistance mutations | 1 year
  * detection of MG resistance mutations macrolide/fluoroquinolone in MG positive samples divided by the total number of MG positive samples
  * detection of MG resistance mutations macrolide/fluoroquinolone in MG positive samples divided by the total number of samples collected

SECONDARY OUTCOMES:
prevalence of CT infection | 1 year
  detection of CT infections in self-collected samples divided by the total number of samples collected
prevalence of NG infection | 1 year
  detection of NG infections in self-collected samples divided by the total number of samples collected
prevalence of syphilis | 1 year
  total number of reported syphilis diagnosis divided by total number of participants tested for syphilis in the clinic
prevalence of HCV infection | 1 year
  total number of reported HCV diagnosis divided by total number of participants tested for HCV in the clinic
prevalence of overall STI | 1 year
  total number of reported STI diagnosis divided by total number of participants tested for STI in the clinic

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong, China, Hong Kong

IPD SHARING:
Plan to Share IPD: No